CLINICAL TRIAL: NCT03412487
Title: Ovarian Histopathology and Laparoscopic Assessment of Premature Ovarian Failure and Its Relation to Thyroid Dysfunction
Brief Title: Ovarian Histopathology and Laparoscopic Assessment of Premature Ovarian Failure
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Cairo University (Other)
Responsible Party: Principal Investigator, Ahmed Maged, professor, Cairo University
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Diagnostic
Other Study IDs: 21
Record Dates: First submitted 2018-01-21; First posted 2018-01-26 (Actual); Last update posted 2018-01-26 (Actual); Status verified 2018-01

CONDITIONS: Premature Ovarian Failure
MeSH Terms: conditions — Primary Ovarian Insufficiency | interventions — Laparoscopy

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- premature ovarian failure (Active Comparator): women under 40 years old with History of oligomenorrhea or amenorrhea for 1 year or more FSH level >20 IU/L at least 2 occasions 4-6 weeks apart (FSH level 20-40 IU/L indicates ovarian insufficiency, while level above 40 IU/L indicates complete failure).
  Interventions: Procedure: laparoscopy
- Control group (Active Comparator): A group of female patients presented with infertility but with regular menses and normal ovarian function (according to history, general examination, gynecological examination and FSH level).
  Interventions: Procedure: laparoscopy

INTERVENTIONS:
Procedure: laparoscopy — under general anesthesia. CO2 pneumoperitoneum, the laparoscope inserted through the umbilicus and a thorough evaluation of the abdominal cavity and pelvis was performed. a grasper was inserted; the utero-ovarian ligament was stabilized with the round biopter will be introduced. The tip of the biopsy instrument was placed on an area of the ovary free of cysts; the hilar area was avoided because it is deficient in small follicles. After correct placement was verified, the inner protecting trocar was removed to expose the sharp leading edge of the round sheath. Gentle circular movements were made cutting through the ovarian cortex to produce a 5-mm disk of 2-3 mm in thickness.

SUMMARY:
25 women with Premature Ovarian Failure who attended Fayoum university hospital gynecology outpatient clinic (case group) and another group of 25 women with normal ovarian function (control group).

*Pelvic laparoscopy and ovarian biopsy will be done ovarian biopsy preparation

For assessment of autoimmune oophoritis, sections were immunostained with anti-LCA (CD45) monoclonal antibody

DETAILED DESCRIPTION:
25 women with Premature Ovarian Failure who attended Fayoum university hospital gynecology outpatient clinic (case group) and another group of 25 women with normal ovarian function (control group).Pelvic laparoscopy and ovarian biopsy To be examined histologically. All procedures were performed under general anesthesia the utero-ovarian ligament was stabilized with the round biopter introduced through the other. The round metal biopter 5 mm in diameter with an inner protective trocar.

The tip of the biopsy instrument was placed on an area of the ovary free of cysts; the hilar area was avoided because it is deficient in small follicles. After correct placement was verified, the inner protecting trocar was removed to expose the sharp leading edge of the round sheath. Gentle circular movements were made cutting through the ovarian cortex to produce a 5-mm disk of 2-3 mm in thickness. The round biopter was removed, and a grasper was introduced to recover the excised tissue.

Ovarian biopsy specimens were fixed in 10% formalin and embedded in paraffin forming tissue blocks. Two sections, 4μ thick were cut from each block. One was stained with routine haematoxylin and eosin (H&E) stain while the other was immunostained with anti-Leukocyte Common Antigen (LCA).

For assessment of autoimmune oophoritis, sections were immunostained with anti-LCA (CD45) monoclonal antibody

ELIGIBILITY:
Inclusion Criteria:

* Woman under age of 40y.

  * Infertility.
  * History of oligomenorrhea or amenorrhea for 1 year or more FSH level >20 IU/L at least 2 occasions 4-6 weeks apart (FSH level 20-40 IU/L indicates ovarian insufficiency, while level above 40 IU/L indicates complete failure).
  * History of thyroid dysfunction, postpartum thyroiditis and or thyroid surgery.
  * Symptoms or signs suggestive of thyroid dysfunction or goiter.
  * Family history of thyroid dysfunction or goiter.
  * Presence of thyroid antibodies or other antibodies.
  * Type 1 Diabetes Mellitus.
  * Prior irradiation to head and neck

Exclusion Criteria:

* Women above 40 yrs.

  * Follicle stimulating hormone (FSH) less than 20mIU/mL
  * Women using hormonal treatement, exposed to radiation to abdomen or pelvis, chemotherapy, or ovarian surgery.

Ages: 20 Years to 40 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Gender Based: Yes
Enrollment: 50 (Estimated)
Dates: Start 2018-01 (Estimated); Primary Completion 2018-12 (Estimated); Study Completion 2019-01 (Estimated)

PRIMARY OUTCOMES:
presence of autoimuune oophoritis | at time of laproscopy procedure
  Autoimmune oophritis was assessed by quantifying LCA positive cells in ovarian stroma as follows:
  [Type text] 0= not convincing.
  1. mild autoimmune oophritis.
  2. moderate autoimmune oophritis.
  3. sever autoimmune oophritis.

CONTACTS AND LOCATIONS:
Overall Officials: Ahmed Maged, MD, Principal Investigator — professor
Locations (1):
- Kasr Alainy medical school, Cairo, Egypt

IPD SHARING:
Plan to Share IPD: Undecided